CLINICAL TRIAL: NCT01462916
Title: Effect of Honey Bee Honey Intake on Children With Chronic Immune Thrombocytopenia
Brief Title: Honey in Chronic Immune Thrombocytopenia
Status: Terminated | Type: Observational
Why Stopped: problem with the candidate (investigator)
Sponsor: mamdouh abdulmaksoud abdulrhman (Other)
Responsible Party: Sponsor-Investigator, mamdouh abdulmaksoud abdulrhman, professor of pediatrics, faculty of medicine, ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: ITP 123
Record Dates: First submitted 2011-10-21; First posted 2011-11-01 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Chronic Thrombocytopenic Purpura
Keywords: honey; mucositis; bee products
MeSH Terms: conditions — Mucositis | interventions — Honey

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- honey, no honey
  Interventions: Dietary Supplement: honey

INTERVENTIONS:
Dietary Supplement: honey — A crossover design (two 12-weeks intervention periods) will be used to measure treatment effects. The subjects will be randomized into two groups (intervention to control [I/C] and control to intervention [C/I] groups). Each study group will have 15 subjects. The subjects in the I/C group will consume 2 ml honey/kg/dose (maximum 50 ml/dose), twice weekly in the first 12-week period (period 1) while the subjects in the C/I group will not receive honey as a Control in period 1. After period 1 the subjects of each group will exchange their protocol for the following 12-week period (period 2).

SUMMARY:
Based on the assumption that honey may have an immunomodulatory effect, the aim of our present study will be to verify whether the intake of honey, as a natural substance, in patients with chronic Immune Thrombocytopenia (ITP) could affect the platelet number and hence could affect the bleeding severity. Thirty patients suffering from chronic ITP will be recruited from the Hematology Clinic of the Pediatric Hospital of Ain Shams University, Cairo, Egypt. The diagnosis of ITP will be based on the presence of isolated thrombocytopenia with a peripheral blood platelet count less than 100 x 109/L, and absence of any obvious initiating and/or underlying cause of the thrombocytopenia. Chronic ITP is defined as ITP for at least 12 months. The age of the patients will range from 5 to 15 years, and they will be of both sexes. This study was approved by the local Ethics Committee of the Pediatric Department of Ain Shams University, and an informed consent to participate in this study will be obtained from at least one parent of each patient. Furthermore, an ascent form will be obtained from each patient above 7 years of age.

DETAILED DESCRIPTION:
Study design:

A crossover design (two 12-weeks intervention periods) will be used to measure treatment effects. The subjects will be randomized into two groups (intervention to control [I/C] and control to intervention [C/I] groups). Each study group will have 15 subjects. The subjects in the I/C group will consume 2 ml honey/kg/dose (maximum 50 ml/dose), twice weekly in the first 12-week period (period 1) while the subjects in the C/I group will not receive honey as a Control in period 1. After period 1 the subjects of each group will exchange their protocol for the following 12-week period (period 2). This design will allow the treatment effects to be measured between the study groups (namely between the different subjects) in the same study period, or period 1, as well as in the same subjects in a crossover comparison of periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic ITP who did not receive any treatment specific for ITP within the past 3 months
2. Who did not receive bee honey or any medication that may affect platelet number or function within the past 3 months and
3. In whom the bleeding severity will range from 1 to 3 (mild to moderate bleeding) according to Buchanan and Adix (2002).

Exclusion Criteria:

1. Grade 4 bleeding severity, according Buchanan and Adix (2002) and
2. Presence of diabetes mellitus.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thirty patients suffering from chronic immune thrombocytopenic purpura (ITP) will be recruited from the Hematology Clinic of the Pediatric Hospital of Ain Shams University,Egypt. The age of the patients will range from 5 to 15 years, and they will be of both sexes.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Bleeding severity | up to 24 weeks
  Bleeding severity will be assessed clinically at least twice weekly and whenever indicated through telephone contact with parents or guardian At least twice weekly for 24 weeks

SECONDARY OUTCOMES:
Platelet count | up to 24 weeks
  Both bleeding severity and platelet count will be assessed at least twice weekly and whenever indicated through telephone contact with parents or guardian At least twice weekly for 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh Abdulrhman, Prof, Principal Investigator — professor; Mohsen El Alfy, prof, Principal Investigator — professor; Abeer Abdulmaksoud, MD, Principal Investigator — Assistant Professor; Abeer Saad, MD, Principal Investigator — Assistant professor; May Said, Principal Investigator — Resident
Locations (1):
- Pediatric Department, Faculty of Medicine, Ain Shams University, Cairo, Egypt

REFERENCES:
- See also: Ain Shams University, Egypt — http://mis2.shams.edu.eg